CLINICAL TRIAL: NCT06310746
Title: A Randomized, Double-Blind, Placebo-Controlled, Single-Dose Escalation Phase I Clinical Study to Assess the Safety, Pharmacokinetics, and Immunogenicity of HLX6018 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HLX6018-FIH101
Record Dates: First submitted 2024-03-07; First posted 2024-03-15 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: IPF

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HLX6018 (Experimental)
  Interventions: Drug: GARP/TGF-β1 monoclonal antibody
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GARP/TGF-β1 monoclonal antibody — It is planned to enroll 8-10 subjects in each of seven dose groups (0.25 mg/kg, 1.0 mg/kg, 4.0 mg/kg, 12 mg/kg, 25 mg/kg, 50 mg/kg, and 70 mg/kg).
  Arms: HLX6018
Drug: Placebo — It is planned to enroll 8-10 subjects in each of seven dose groups (0.25 mg/kg, 1.0 mg/kg, 4.0 mg/kg, 12 mg/kg, 25 mg/kg, 50 mg/kg, and 70 mg/kg).
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the safety, PK, and immunogenicity of a single intravenous administration of HLX6018 in healthy subjects, based on the preliminary efficacy and safety established through in vitro and in vivo experiments.

This is a randomized, double-blind, placebo-controlled study with single dose escalation design to assess the safety, PK, and immunogenicity of HLX6018 in healthy subjects. It is planned to enroll 8-10 subjects in each of seven dose groups (0.25 mg/kg, 1.0 mg/kg, 4.0 mg/kg, 12 mg/kg, 25 mg/kg, 50 mg/kg, and 70 mg/kg). This is the first-in-human study of the investigational product.

ELIGIBILITY:
Inclusion Criteria:

1. Fully informed about the nature, significance, potential inconveniences, and associated risks of the study prior to enrollment. Comprehend the study's procedures and methodology, agree to follow the clinical study protocol, and give voluntary written informed consent;
2. 18-55 years old, including the boundary value, male or female;
3. Body weight: 45-85 kg for females and 50-85 kg for males, including the boundary value; body mass index (BMI): 18.0-28.0 kg/m2 , including the boundary value, (BMI = body weight (kg)/body height2 (m2));
4. Subjects, including males, must have no childbearing plan and take effective contraceptive measures from the time of informed consent to 6 months after the administration of the study drug.
5. Physical examinations and vital signs should be normal or abnormal without clinical significance.

Exclusion Criteria:

1. Any clinically significant laboratory test abnormalities or, within 12 months before screening, any other clinically significant clinical findings indicative of diseases, including but not limited to gastrointestinal, renal, hepatic, neurological, hematological, endocrine, oncological, pulmonary, immunological, psychiatric, or cardiovascular conditions;
2. Donation/loss of ≥ 450 mL of blood or receipt of blood transfusion or use of blood products within 3 months prior to screening, or planning to donate blood during the study or within 1 month after the end of the study;
3. Patients with severe trauma or major surgery within 3 months before screening, or planning to undergo surgery during the study;
4. Patients who smoke more than 5 cigarettes per day in the 3 months before screening;
5. History of drug abuse or addiction or alcohol abuse (14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of spirits, or 100 mL of wine);

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2024-04-23 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
The number of subjects experiencing adverse events (AEs) and serious adverse events (SAEs) | 0 to Day 99
  Safety evaluation

SECONDARY OUTCOMES:
AUC0-inf | 0 to Day 99
  Area under the serum concentration-time curve
Cmax | 0 to Day 99
  Peak concentration
Tmax | 0 to Day 99
  Time to reach peak concentration
T1/2 | 0 to Day 99
  Terminal elimination half-life
CL | 0 to Day 99
  Clearance
λz | 0 to Day 99
  Terminal elimination rate constant

CONTACTS AND LOCATIONS:
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No